CLINICAL TRIAL: NCT02187367
Title: Phase 3 Open-label, Multicentre, Randomised Trial to Establish Safety & Efficacy of an EGF Cancer Vaccine in Inoperable, Stage IV Biomarker Positive,Wild Type EGF-R NSCLC Patients Eligible to Receive Standard Treatment and Supportive Care
Brief Title: Safety & Efficacy Study of EGF Cancer Vaccine to Treat Stage IV Biomarker Positive, Wild Type EGF-R NSCLC Patients
Acronym: EGF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on slow recruitment and new emerging drug combinations
Sponsor: Bioven Europe (Industry)
Responsible Party: Sponsor
Organization: Bioven Sdn. Bhd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BV-NSCLC-002; 2013-005335-25 (EudraCT Number)
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGF Vaccine (Experimental): Patients in this arm will receive a low dose of cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51
  Interventions: Biological: EGF Vaccine
- Best Supportive Care (No Intervention): Patients in this arm will receive best supportive care

INTERVENTIONS:
Biological: EGF Vaccine — 1.2mL of conjugate-adjuvant mix injection at four sites during the Post First-Line Chemotherapy. Reduced dose of injection at two sites during the Pre-Progression Phase.
  Other Names: Cyclophosphamide and the recombinant human rEGF-P64K/Montanide ISA 51
  Arms: EGF Vaccine

SUMMARY:
The vaccine contains humanized recombinant antigen (EGF - Epithelial Growth Factor) and an adjuvant. The antibodies induced by vaccination will react with circulating EGF leading to removal of EGF from the circulation. As a result, binding to its target EGF-Receptor is prevented. Blocking of EGF-Receptor is preventing activation and stimulation of proliferation of tumour cell. A Phase 3 clinical trial on the EGF vaccine is ongoing in Cuba. The result from previous studies demonstrated positive correlation between extended survival and immune response against the vaccination in the late-stage NSCLC patients' age below 60 with improved quality of life. The purpose of this international Phase 3 trial is to determine whether the recombinant human EGF cancer vaccine is safe, immunogenic and effective in the treatment of stage IV NSCLC patients who are positive in the selective EGF biomarker and wild type EGF-Receptor compared to standard treatment and supportive care.

ELIGIBILITY:
Inclusion Criteria:

1. Are aged 18 or older.
2. Have serum EGF concentration >250 pg/ml determined from sample taken at screening.
3. Have wild type EGF-R sequence.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Have adequate bone marrow, liver and renal function, as assessed by the Investigator. A sample taken at Screening should confirm that:

   * White blood cell (WBC) count ≥ 3000 per µL
   * Platelet count ≥ 100,000 per µL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) (or ≤ 5 x ULN when liver metastases are present)
   * Total bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
6. Have histologically and/or cytologically confirmed diagnosis of NSCLC, corresponding to locally and regionally advanced inoperable disease (Stage IV [as defined by the American Joint Committee on Cancer staging system- TNM 7th edition 2010]) excluding brain metastases.
7. Are eligible to receive first-line chemotherapy (without concurrent radiotherapy to thorax measurable lesions or consolidation radiotherapy).
8. Agree to use double-barrier contraception (males and females alike [if applicable]). A negative pregnancy test must be documented at Screening for females of childbearing potential.

   Note: Females of childbearing potential are defined as those women with less than 2 years after last menstruation and not surgically sterile, while post-menopausal refers to those women with at least 2 years from last menstruation.
9. Have signed a voluntary written informed consent form (ICF). Patients should be cooperative, willing and able to participate and adhere to the Protocol requirements, including their availability for the follow-up.

Exclusion Criteria:

1. Patient has no measurable disease (as defined by RECIST Criteria, version 1.1).
2. Patient has EGF-R mutation.
3. Patient has EGF serum concentration below required threshold.
4. Patient is a candidate for concurrent chemo-radiotherapy or post chemo thoracic radiotherapy.
5. Patient has a history of known or suspected central nervous system (CNS) metastases.
6. Patient has a history of primary malignancy (except resected non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix), unless in complete remission and off all chemotherapy and/or radiotherapy for that disease for a minimum of 5 years. Any palliative radiotherapy to alleviate pain in bone metastases is permitted.
7. Patient is taking immunosuppressant drugs such as azathioprine, tacrolimus, cyclosporine, etc. Use is not permitted within 1 month before Screening.
8. Patient is taking any other immunotherapy.
9. Patient has primary or secondary immunodeficiencies (e.g. documented Human Immunodeficiency Virus [HIV]).
10. Patient has autoimmune disease.
11. Patient has undergone splenectomy.
12. Patient is taking oral, intramuscular or intravenous corticosteroids. Use is not permitted within 1 month before Screening. Inhaled corticosteroids to treat respiratory insufficiency (e.g. chronic obstructive pulmonary disease [COPD]), or topical steroids are permitted.
13. Patient has neurotoxicity (Grade ≥2).
14. Patient has diarrhoea (Grade ≥2).
15. Patient has received other vaccines (with the exception of the influenza vaccine), within 1 month before Screening.
16. Patient has a history of any severe or life-threatening hypersensitivity reaction.
17. Patient has an unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal and metabolic disease).
18. Patient has recent history (within 6 months before Screening) of chronic alcohol or drug abuse which may compromise the patient's safety or ability to participate in study activities.
19. Patient has a history of psychiatric disorder that prevents patients from providing informed consent or following Protocol instructions.
20. Patient is currently enrolled in an investigational device or drug trial, or <1 month since completing an investigational device or drug trial.
21. Female patients who are pregnant or lactating.
22. Patient has any other factor that in the opinion of the Investigator (or designee) would make the patient unsafe or unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Each patient will be followed till death occurs within study time frame of 3 years
  To assess overall survival (OS) of an EGF cancer vaccine in inoperable, stage IV biomarker positive, wild type EGF-R, NSCLC patients compared to the control group receiving best treatment and supportive care. OS is defined as the time from randomisation to death due to any cause.

SECONDARY OUTCOMES:
Safety of EGF Cancer Vaccine as assessed by Adverse Events (AEs) | Each patient will be followed till death occurs within study time frame of 3 years
  To assess the frequency and number of patients develop AEs, related AEs, serious AEs (SAEs) and AEs leading to withdrawal or death
Progression-Free Survival (PFS) | Each patient will be followed till objective tumour progression or death (whichever occurs first) within time frame of study of 3 years
  Progression parameters include radiological or clinical progression, withdrawal due to progression, and death due to any cause.
Survival Rate | Each patient will be followed at 12 and 24 months after randomization
  To assess the percentage of patients that are alive at 12 months and 24 months in EGF cancer vaccine study group compared to control group.
Time to Progression (TTP) | Each patient will be followed till observed tumour progression within study time frame of 3 years
  To assess Time to Progression (TTP) from the time of randomisation to first documented disease progression of EGF cancer vaccine study group patients compared to control group.
Response Rate (RECIST criteria) | Each patients will be followed till death occurs within study time frame of 3 years
  To assess the percentage of patients with a complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria Version 1.1.
Safety of EGF Cancer Vaccine by Laboratory Assessment | Each patients will be followed till death occurs within study time frame of 3 years
  To assess haematology, biochemistry and urinalysis parameters
Safety of EGF Cancer Vaccine assessed by Vital Signs | Each patients will be followed till death occurs within study time frame of 3 years
  To assess systolic and diastolic blood pressure, body temperature and pulse rate
Safety of EGF Cancer Vaccine as assessed by Physical Examination | Each patient will be followed till death occurs within study time frame of 3 years
  To assess eyes, neurological and cardiovascular systems, lungs, abdomen, and any other areas with signs and symptoms of disease, and of the head, neck, ears, nose, mouth, throat, thyroid, lymph nodes and extremities
Quality of Life (QoL) | Each patient will be followed till death occurs within study time frame of 3 years
  To assess the general physical health of patients with a 36-item, short-form health survey until disease progression

OTHER OUTCOMES:
Pharmacodynamics (PD) of EGF Cancer Vaccine assessed by Immune Responses | Each patients will be followed till death within study time frame of 3 years
  To assess the serum EGF concentration and anti-EGF antibody titers with response before and after to the study treatment
Efficacy assessed by KRAS and ALK rearrangements | At time of screening
  For the analysis of oncogenes Kirsten rat sarcoma (KRAS) and anaplastic lymphoma kinase (ALK), a formalin-fixed, paraffin embedded (FFPE) sample of the biopsy tumour tissue, ideally taken from biopsy obtained at disease diagnosis will be prepared and shipped for central analysis

CONTACTS AND LOCATIONS:
Overall Officials: Libor Havel, Dr., Principal Investigator — Thomayerova nemocnice, Czech Republic
Locations (51):
- Bulgaria (2):
  - "Multiprofile Hospital for Active Treatment (MHAT)-Dobrich" AD, Dobrich
  - MHAT for Women's Health-Nadezhda"OOD, Sofia
- Czechia (3):
  - Nemocnice Na Pleši s.r.o. Oddelení klinické onkologie a radioterapie, Nová Ves pod Pleší
  - Pardubická krajská nemocnice, a.s.c, Pardubice
  - Thomayerova nemocnice, Prague
- Georgia (8):
  - Cancer Center of Adjara, Batumi
  - Clinic Health House, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - JSC, Maritime Hospital, Tbilisi
  - JSC, Neo Medi, Tbilisi
  - LTD, High Technology Medical Centre, University Clinic, Tbilisi
  - LTD, Medulla - Chemotherapy and Immunotherapy Clinic, Tbilisi
  - Research Institute Of Clinical Medicine, Tbilisi
- Germany (9):
  - Universitätsklinikum Halle (Saale) Klinik und Poliklinik fuer Innere Medizin, Halle, Saale
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Kliniken der Stadt Köln GmbH, Cologne
  - KRH Klinikum Siloah Hannover - Oststadt, Hanover
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel
  - Universitätsklinikum Leipzig - AöR, Leipzig
  - LMU-München, München
  - Mühlen-Apotheke, Oststeinbek
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Sarawak General Hospital, Kuching
  - Mahkota Medical Center, Malacca
  - Hospital Pulau Pinang, Pulau Pinang
- Philippines (7):
  - Perpetual Succour Hospital, Lahug, Cebu City
  - Makati Medical Center, Makati, Manila
  - The Medical City, Pasig, National Capital Region
  - Lung Center of the Philippines, Quezon City, National Capital Region
  - Davao Doctors hospital, Davao City
  - Cancer Research Center, Manila
  - Philippine General Hospital, Manila
- Poland (2):
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Szpital Specjalistyczny w Prabutach, Prabuty
- Romania (3):
  - Centrul de Oncologie "Sf. Nectarie", Craiova
  - S.C. R.T.C. Radiology Therapeutic Center S.R.L., Otopeni
  - SC Oncomed SRL, Târgu Mureş
- Spain (5):
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jimenez Díaz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Thailand (5):
  - Lopburi Cancer Hospital, Mueang, Changwat Lop Buri
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Bangkok Hospital Chiang Mai, Bangkok
  - Lampang Cancer Hospital, Lampang
  - Buddhachinaraj Hospital, Phitsanulok
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Nottingham University Hospitals, Nottingham
  - University Hospital Southampton NHS Trust, Southampton